CLINICAL TRIAL: NCT00470223
Title: OS2006 : Protocole de Traitement Des ostéosarcomes de l'Enfant, de l'Adolescent et de l'Adulte Comportant
Brief Title: Combined Chemotherapy With or Without Zoledronic Acid for Patients With Osteosarcoma
Acronym: OS2006
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: UNICANCER (Other)
Collaborators: Novartis (Industry); Chugai Pharmaceutical (Industry); National Cancer Institute, France (Other Government); SFCE (Unknown); Ligue contre le cancer, France (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Sarcome 09/0603; UNICANCER-SARCOME-09-0603 (Other: UNICANCER); 2006-003377-27 (EudraCT Number)
Record Dates: First submitted 2007-05-03; First posted 2007-05-07 (Estimated); Last update posted 2025-06-08 (Actual); Status verified 2025-05

CONDITIONS: Sarcoma
Keywords: localized osteosarcoma; metastatic osteosarcoma
MeSH Terms: conditions — Sarcoma; Osteosarcoma | interventions — Cisplatin; Doxorubicin; Etoposide; Ifosfamide; Methotrexate; Zoledronic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Chemotherapy + zoledronic acid (Experimental)
  Interventions: Drug: cisplatin; Drug: doxorubicin hydrochloride; Drug: etoposide; Drug: ifosfamide; Drug: methotrexate; Drug: zoledronic acid; Procedure: conventional surgery
- chemotherapy (Active Comparator)
  Interventions: Drug: cisplatin; Drug: doxorubicin hydrochloride; Drug: etoposide; Drug: ifosfamide; Drug: methotrexate; Procedure: conventional surgery

INTERVENTIONS:
Drug: cisplatin
Drug: doxorubicin hydrochloride
Drug: etoposide
Drug: ifosfamide
Drug: methotrexate
Drug: zoledronic acid
  Arms: Chemotherapy + zoledronic acid
Procedure: conventional surgery

SUMMARY:
RATIONALE: Drugs used in chemotherapy work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving more than one drug (combination chemotherapy) may kill more tumor cells. Zoledronic acid may stop the growth of tumor cells in bone. Giving chemotherapy with or without zoledronic acid before surgery may make the tumor smaller and reduce the amount of normal tissue that needs to be removed. Giving these treatments after surgery may kill any tumor cells that remain after surgery. It is not yet known whether giving combination chemotherapy together with zoledronic acid is more effective than combination chemotherapy alone in treating osteosarcoma.

PURPOSE: This randomized phase III trial is studying combination chemotherapy and zoledronic acid to see how well they work compared with combination chemotherapy alone in treating patients with osteosarcoma.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Compare the progression-free survival of patients with osteosarcoma treated with combination chemotherapy with or without zoledronic acid.

Secondary

* Compare the overall survival of patients treated with these regimens.
* Compare the percentage of patients with a good histologic response.
* Compare the long and short term toxicity of these regimens in these patients.
* Compare the quality of life of patients treated with these regimens.

OUTLINE: This is a randomized, multicenter study. Patients are stratified according to age (< 18 years vs 18-25 years vs > 25 years), risk group (nonmetastatic or resectable vs metastatic or unresectable), and treatment center. Patients receive either methotrexate-based chemotherapy or doxorubicin hydrochloride-based chemotherapy according to age.

* Methotrexate-based chemotherapy (patients ≤ 25 years of age): Patients are randomized to 1 of 2 treatment arms.

  * Arm I: Patients receive methotrexate IV in weeks 1-3, 7, 8, 12, and 13 and etoposide IV and ifosfamide IV in weeks 4 and 9.
  * Arm II: Patients receive methotrexate, etoposide, and ifosfamide as in arm I. Patients also receive zoledronic acid IV in weeks 1, 5, 9, and 13.

All patients undergo surgery in week 14. After surgery, patients are assigned to 1 of 2 groups for further treatment, based on histological response.

* Good responders (< 10% viable cells): Patients are randomized to 1 of 2 treatment arms.

  * Arm I: Patients receive methotrexate IV in weeks 1-3, 7-9, 13-15, and 19-21 and etoposide IV in weeks 4 and 10. Patients also receive ifosfamide IV in weeks 4, 10, and 16.
  * Arm II: Patients receive methotrexate, etoposide, and ifosfamide as in arm I. Patients also receive zoledronic acid IV in weeks 3, 7, 11, 15, 19, and 23.
* Bad responders (> 10% viable cells): Patients are randomized to 1 of 2 treatment arms.

  * Arm I: Patients receive methotrexate IV in weeks 1, 5, 9, 13, and 17 and doxorubicin hydrochloride IV and cisplatin IV in weeks 2, 6, 10, 14, and 18.
  * Arm II: Patients receive methotrexate, doxorubicin hydrochloride, and cisplatin as in arm I. Patients also receive zoledronic acid IV as in arm II (good responders).

    * Doxorubicin hydrochloride-based chemotherapy (patients ≥ 18 years of age): Patients are randomized to 1 of 2 treatment arms.
* Arm I: Patients receive doxorubicin hydrochloride IV and ifosfamide hydrochloride IV in weeks 1, 4, 7, 10, and 13 and cisplatin IV in weeks 1, 7, and 13.
* Arm II: Patients receive doxorubicin hydrochloride, ifosfamide, and cisplatin as in arm I. Patients also receive zoledronic acid IV in weeks 1, 5, 9, and 13.

All patients undergo surgery in week 16. After surgery, patients are assigned to 1 of 2 groups for further treatment, based on histological response.

* Good responders (< 10% viable cells): Patients are randomized to 1 of 2 treatment arms.

  * Arm I: Patients receive doxorubicin hydrochloride IV in weeks 1 and 7 and ifosfamide IV in weeks 1, 4, 7, and 10.
  * Arm II: Patients receive doxorubicin hydrochloride and ifosfamide as in arm I. Patients also receive zoledronic acid IV in weeks 1, 5, 9, 13, 17, and 21.
* Bad responders (> 10% viable cells):

  * Arm I: Patients receive etoposide IV and ifosfamide IV in weeks 1, 4, 7, 10, and 13.
  * Arm II: Patients receive etoposide and ifosfamide as in arm I. Patients also receive zoledronic acid as in arm II (good responders).

PROJECTED ACCRUAL: A total of 440 patients will be accrued for this study.

ELIGIBILITY:
Inclusion Criteria

* Histologically confirmed high-grade osteosarcoma
* Bilirubin ≤ 2 times upper limit of normal
* No medical condition that would preclude study treatment
* Not pregnant or nursing
* Fertile patients must use effective contraception
* Shortening fraction ≥ 28%
* LVEF ≥ 50%
* Glomerular filtration rate ≥ 70mL/min
* No recent dental problem, including infection, traumatization, or surgery

Exclusion Criteria

* Low-grade osteosarcoma
* Small cell osteosarcoma
* Maxillary osteosarcoma
* Primary resected osteosarcoma
* Osteosarcoma with multiple metastases for which complete removal is not feasible even after shrinkage with chemotherapy
* Extra-osseous osteosarcoma
* Any prior osteonecrosis of the maxilla
* No prior chemotherapy or radiotherapy

Ages: 5 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 318 (Actual)
Dates: Start 2007-03 (Actual); Primary Completion 2015-12 (Actual); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Event-free survival | 3 years

SECONDARY OUTCOMES:
Overall survival | 10 years
Percentage of good responders | at the time of the surgery
Short term and long term toxicity | 10 years

CONTACTS AND LOCATIONS:
Overall Officials: Laurence Brugieres, MD, Study Chair — Gustave Roussy, Cancer Campus, Grand Paris
Locations (37):
- France (37):
  - Centre Paul Papin, Angers
  - Institut Gustave Roussy, Angers
  - Centre Hospitalier Regional de Besancon - Hopital Jean Minjoz, Besançon
  - CHR de Besancon - Hopital Saint-Jacques, Besançon
  - Institut Bergonie, Bordeaux
  - CHU Hopital A. Morvan, Brest
  - CHU de Caen, Caen
  - Centre Regional Francois Baclesse, Caen
  - CHR Clermont Ferrand, Hotel Dieu, Clermont-Ferrand
  - Centre Jean Perrin, Clermont-Ferrand
  - Centre de Lutte Contre le Cancer Georges-Francois Leclerc, Dijon
  - Centre Hospitalier Universitaire de Dijon, Dijon
  - CHU de Grenoble - Hopital Michallon, Grenoble
  - Centre Oscar Lambret, Lille
  - Centre Leon Berard, Lyon
  - Hopital Edouard Herriot - Lyon, Lyon
  - Marseille Institute of Cancer - Institut J. Paoli and I. Calmettes, Marseille
  - CHU de la Timone, Marseille
  - Hopital d'Enfants de la Timone, Marseille
  - CHU Nord, Marseille
  - Hopital Arnaud de Villeneuve, Montpellier
  - Centre Regional de Lutte Contre le Cancer - Centre Val d'Aurelle, Montpellier
  - Centre Antoine Lacassagne, Nice
  - Hopital de l'Archet CHU de Nice, Nice
  - Institut Curie Hopital, Paris
  - Hopital Jean Bernard, Poitiers
  - Centre Eugene Marquis, Rennes
  - Hopital Charles Nicolle, Rouen
  - Centre Henri Becquerel, Rouen
  - Centre Regional Rene Gauducheau, Saint-Herblain
  - Institut de Cancerologie de la Loire, Saint-Priest-en-Jarez
  - Hopitaux Universitaire de Strasbourg, Strasbourg
  - Hopital Universitaire Hautepierre, Strasbourg
  - Hopital des Enfants, Toulouse
  - C.H. Bastien de Clocheville, Tours
  - CHRU de Tours - Hopital Trousseau, Tours
  - Centre Alexis Vautrin, Vandœuvre-lès-Nancy

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared at an individual level, they will be part of the study database including all enrolled patients.

REFERENCES:
- [Derived] Hattinger CM, Patrizio MP, Magagnoli F, Luppi S, Serra M. An update on emerging drugs in osteosarcoma: towards tailored therapies? Expert Opin Emerg Drugs. 2019 Sep;24(3):153-171. doi: 10.1080/14728214.2019.1654455. Epub 2019 Aug 14. PMID 31401903
- [Derived] Lui G, Treluyer JM, Fresneau B, Piperno-Neumann S, Gaspar N, Corradini N, Gentet JC, Marec Berard P, Laurence V, Schneider P, Entz-Werle N, Pacquement H, Millot F, Taque S, Freycon C, Lervat C, Le Deley MC, Mahier Ait Oukhatar C, Brugieres L, Le Teuff G, Bouazza N; Sarcoma Group of UNICANCER. A Pharmacokinetic and Pharmacogenetic Analysis of Osteosarcoma Patients Treated With High-Dose Methotrexate: Data From the OS2006/Sarcoma-09 Trial. J Clin Pharmacol. 2018 Dec;58(12):1541-1549. doi: 10.1002/jcph.1252. Epub 2018 May 23. PMID 29791011
- [Derived] Tabone MD, Brugieres L, Piperno-Neumann S, Selva MA, Marec-Berard P, Pacquement H, Lervat C, Corradini N, Gentet JC, Couderc R, Chevance A, Mahier-Ait Oukhatar C, Entz-Werle N, Blay JY, Le Deley MC. Prognostic impact of blood and urinary angiogenic factor levels at diagnosis and during treatment in patients with osteosarcoma: a prospective study. BMC Cancer. 2017 Jun 15;17(1):419. doi: 10.1186/s12885-017-3409-z. PMID 28619014
- [Derived] Piperno-Neumann S, Le Deley MC, Redini F, Pacquement H, Marec-Berard P, Petit P, Brisse H, Lervat C, Gentet JC, Entz-Werle N, Italiano A, Corradini N, Bompas E, Penel N, Tabone MD, Gomez-Brouchet A, Guinebretiere JM, Mascard E, Gouin F, Chevance A, Bonnet N, Blay JY, Brugieres L; Sarcoma Group of UNICANCER; French Society of Pediatric Oncology (SFCE); French Sarcoma Group (GSF-GETO). Zoledronate in combination with chemotherapy and surgery to treat osteosarcoma (OS2006): a randomised, multicentre, open-label, phase 3 trial. Lancet Oncol. 2016 Aug;17(8):1070-1080. doi: 10.1016/S1470-2045(16)30096-1. Epub 2016 Jun 17. PMID 27324280